CLINICAL TRIAL: NCT07257913
Title: Impact of Dairy Integration Into Canadian Food Guide on Gut Health
Acronym: GutMilk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alain Veilleux, Full professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-569
Record Dates: First submitted 2025-09-22; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Gut Epithelial Permeability; Gut Microbiota Composition and Diversity; Gut and Circulating Inflammatory Markers; Milk and Digestion
Keywords: Milk consumption; Gut epithelial permeability; Inflammation; Gut microbiota
MeSH Terms: conditions — Inflammation | interventions — Milk; Cultured Milk Products; Soy Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Milk (Experimental): - Consumption of milk 3 times per day during 9 days alongside CFG diet, following a 4 day control diet
  Interventions: Other: Milk; Other: Fermented milk; Other: Soy beverage
- Fermented milk (Experimental): - Consumption of fermented milk 3 times per day during 9 days alongside CFG diet, following a 4 day control diet
  Interventions: Other: Milk; Other: Fermented milk; Other: Soy beverage
- Soy beverage (Experimental): - Consumption of a soy beverage 3 times per day during 9 days alongside CFG diet, following a 4 day control diet
  Interventions: Other: Milk; Other: Fermented milk; Other: Soy beverage

INTERVENTIONS:
Other: Milk — Consumption of 1 cup milk 3 times per day during 9 days alongside CFG diet
Other: Fermented milk — Consumption of fermented milk 3 times per day during 9 days alongside CFG diet
Other: Soy beverage — Consumption of a soy beverage 3 times per day during 9 days alongside CFG diet

SUMMARY:
The primary objective is to investigate the impact of milk, fermented milk, and soy beverages, incorporated in a diet reflecting adherence to Canadian food guide recommendations on food choices on gut microbiota in middle-aged adults (45-65 years) with abdominal obesity and slightly deteriorated lipids and/or glucose profile. The study aims to discern whether the integration of soy beverages (control), milk, and fermented milk within the CFG diet contributes to distinct gut outcomes and alterations in gut health. We hypothesized that milk and fermented milk will further promote beneficial changes in gut health parameters including gut microbiota composition, trans-epithelial permeability, and inflammation, relative to soy beverages.

DETAILED DESCRIPTION:
Single-blinded crossover RCT to test the impact of integrating dairy (i.e., milk and fermented milk) into the Canadian Food Guide (CFG) diet on gut health, in fully controlled dietary settings. The trial will include mid-age women and men with abdominal obesity and slightly deteriorated metabolic profile (n=20). The trial will feature 3 controlled-feeding phases (14 days), allocated in a random order and separated by free-uncontrolled feeding washout periods (14-28 days). Each dietary intervention phase will be initiated by a Run-in full-feeding period (4 days), to standardize participants' dietary intakes, and immediately followed by one of the 3 dietary interventions (9 days) reflecting adherence to the CFG recommendation (9 days, CFG-Diet) incorporating either soy beverages (Control), milk, or non-effervescent fermented milk.

This approach was shown to be highly informative in deciphering the interaction between diet and the gut microbiota in previous work. It will be able to assess how integrating dairy (i.e., milk and fermented milk) into the Canadian Food Guide (CFG) diet promptly modulates gut health parameters (i.e. gut microbiota composition, inflammatory states, and gut permeability) in the context of obesity and metabolic complications, relative to a plant-based alternative. The fully controlled dietary setting of this study design will provide precise intakes of foods and bioactive nutrients, which will enable us to comprehensively assess the impact of dairies on gut health.

The trial will include 10 women and 10 men with abdominal obesity and slightly deteriorated metabolic profile.

Diet sequence allocation will be randomized with a sex-specific stratification. The study will be single-blinded, such as participants will not be informed of the precise nature of the diet sequence.

TRIAL INTERVENTION PHASES (3 X 14 DAYS)

During each intervention phases, all meals and foods will be provided to ensure optimal diet control. Each intervention phases will follow this sequence:

* Day 0: Initiation of the run-in full-feeding period (4 days) to standardize participants' dietary intakes.
* Day 4: Baseline sampling and data collection.
* Day 4: Initiation of the CFG dietary intervention (10 days) incorporating either soy beverages (Control), milk, or non-effervescent fermented milk.
* Day 6: Post-intervention (+2 days) sampling and data collection.
* Day 13: Post-intervention (+9 days) sampling and data collection. End of the intervention phases.

ELIGIBILITY:
Inclusion Criteria:

* IMC < 45
* Waist circumference > 80 cm (Women) or 94 cm (men)

Exclusion Criteria:

* History of diabetes (types 1 and 2), CVD, enteropathy, immune diseases or bariatric surgery
* Cancer (diagnostic and/or treatment) during the last 5 years
* Antibiotic consumption during the last 3 months
* Active smoking or cannabis consumption
* Lactose intolerance or allergy, any allergies to foods given in the intervention phases
* Irregular defecation patterns
* Pregnancy/lactation
* Inability to speak French

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Gut epithelial permeability | This outcome will be measured on the last day (day 13) of each intervention phase.
  Post-intervention lactulose/mannitol ratio by LCMS, 0-5 hours after ingestion of the non-metabolizable sugar

SECONDARY OUTCOMES:
Gut inflammatory markers | Samples will be collected on days 6 and 13 of each intervention phase.
  Fecal calprotectin levels by ELISA
Perceived gut symptoms | Gastrointestinal symptoms questionnaire is administered on days 0, 4 and 13.
  Perception gastrointestinal symptoms questionnaires
Whole gut transit time | At days 1, 4 and 11.
  Whole gut transit time (h) by the Blue poop challenge

CONTACTS AND LOCATIONS:
Overall Officials: Alain Veilleux, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication